CLINICAL TRIAL: NCT06627920
Title: Validation of a Smartwatch for Blood Pressure Measurement
Brief Title: Validation of a Smartwatch for Blood Pressure Monitoring
Acronym: SmartBP
Status: Completed | Type: Observational
Sponsor: European University Miguel de Cervantes (Other)
Collaborators: Valladolid University Clinical Hospital. Cardiology Department. (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI-DOC007_SmartBP
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure; Heart Rate; Oxygen Saturation
Keywords: cardiovascular health; wearable devices; blood pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Descriptive: A single population is used to estimate blood pressure, heart rate and oxygen saturation in order to study and validate the use of the KC08 smartwatch.
  Interventions: Device: Use of the KC08 smartwatch, Beurer PO30 and Omron M7 BP monitor.

INTERVENTIONS:
Device: Use of the KC08 smartwatch, Beurer PO30 and Omron M7 BP monitor. — Use of the KC08 smartwatch, Beurer PO30 and Omron M7 BP monitor to estimate blood pressure, heart rate and oxygen saturation.

SUMMARY:
Accurate measurement of blood pressure is essential for the assessment of cardiovascular health and the prevention of cardiovascular disease. Smartwatches have emerged as a promising option for continuous monitoring of blood pressure outside the clinical setting. This study aims to validate the use of the smartwatch KC08 for blood pressure measurement, which is a cost-effective and convenient alternative for blood pressure measurement. A cross-sectional study will be conducted with participants aged greater than or equal to18 years. The measurements of blood pressure, heart rate and oxygen saturation will be performed with the smartwatch KC08, the Beurer PO30 pulse oximeter and the Omron M7 BP monitor. The statistical analysis will evaluate the reliability of the devices and compare the measurements of the two devices using different statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years old and able to understand the informed consent.

Exclusion Criteria:

* A difference of ≥20 mmHg in systolic and/or diastolic blood pressure between both arms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Observational cross-sectional study with participants at least 18 years of age. Participants will be recruited from the European University Miguel de Cervantes. Once the protocol has been explained and the informed consent has been signed, measurements will be taken.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Diastolic and systolic blood pressure | 5 minutes rest; 5 minutes safety BP measurements of both arms; 30 minutes BP measurements (10 measurements in total)
  For BP measurement, an Omron M7 automatic blood pressure monitor (Omron Healthcare Co., Ltd., Kyoto, Japan) and a KC08 smartwatch (Mediatek Inc., Hsinchu, Taiwan) will be used. The participant should sit in a comfortable chair with lumbar support for at least 5 minutes prior to the measurement. The participant will be asked to place both feet flat on the floor, without crossing the legs, and rest the arm with the cuff on a table at chest level, palm up. Ensuring that the cuff is properly adjusted but not too tight and in contact with bare skin, the blood pressure will be measured. During this process, the subject should refrain from talking to ensure an accurate and reliable reading. The values obtained will be recorded according to standard blood pressure measurement procedures. 10 measurements separated by 1 minute will be taken with each device. The BP results will be recorded in mmHg.
Heart rate | 30 minutes (10 measurements in total)
  An Omron M7 automatic blood pressure monitor (Omron Healthcare Co., Ltd., Kyoto, Japan), a Beuer PO30 pulse oximeter and a KC08 smartwatch (Mediatek Inc., Hsinchu, Taiwan) will be used. Heart rate will be recorded while blood pressure measurements are being recorded.
  10 measurements separated by 1 minute will be taken with each device. The heart rate results will be recorded in beats per minute (bpm).
Peripheral oxygen saturation | 30 minutes (10 measurements in total)
  A Beurer PO30 pulse oximeter (Beurer GmbH, Mittelstand, Germany) and a KC08 smartwatch (Mediatek Inc., Hsinchu, Taiwan) will be used. 10 measurements separated by 1 minute will be taken with each device. The peripheral oxygen saturation results will be recorded in percentage of hemoglobin saturation.
Physical activity levels | 2 minutes
  Participants' physical activity levels will be assessed using the International Physical Activity Questionnaire (IPAQ). This questionnaire consists of 7 questions that will help us stratify physical activity levels.
  It is used as a descriptive measure of the users and a possible confounding factor. It takes approximately 2 minutes to complete the questionnaire and we do it in the initial interview, before starting with the measurements of BP, heart rate and peripheral oxygen saturation.

CONTACTS AND LOCATIONS:
Locations (1):
- European University Miguel de Cervantes, Valladolid, Castille and León, Spain

REFERENCES:
- [Background] Jose AP, Awasthi A, Kondal D, Kapoor M, Roy A, Prabhakaran D. Impact of repeated blood pressure measurement on blood pressure categorization in a population-based study from India. J Hum Hypertens. 2019 Aug;33(8):594-601. doi: 10.1038/s41371-019-0200-4. Epub 2019 Apr 12. PMID 30979950
- [Background] Boateng EB, Ampofo AG. A glimpse into the future: modelling global prevalence of hypertension. BMC Public Health. 2023 Oct 3;23(1):1906. doi: 10.1186/s12889-023-16662-z. PMID 37789258
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] Konstantinidis D, Iliakis P, Tatakis F, Thomopoulos K, Dimitriadis K, Tousoulis D, Tsioufis K. Wearable blood pressure measurement devices and new approaches in hypertension management: the digital era. J Hum Hypertens. 2022 Nov;36(11):945-951. doi: 10.1038/s41371-022-00675-z. Epub 2022 Mar 23. PMID 35322181
- [Background] Bradley CK, Shimbo D, Colburn DA, Pugliese DN, Padwal R, Sia SK, Anstey DE. Cuffless Blood Pressure Devices. Am J Hypertens. 2022 May 10;35(5):380-387. doi: 10.1093/ajh/hpac017. PMID 35136906
- [Background] Yi L, Lv ZH, Hu SY, Liu YQ, Yan JB, Zhang H, Li HB, Chen Q, Li YY, Jiang YF, Zhou H, Li MD, Chen RD, Li XL, Zhou SS, Chen YD. Validating the accuracy of a multifunctional smartwatch sphygmomanometer to monitor blood pressure. J Geriatr Cardiol. 2022 Nov 28;19(11):843-852. doi: 10.11909/j.issn.1671-5411.2022.11.004. PMID 36561062
- [Background] Moon JH, Kang MK, Choi CE, Min J, Lee HY, Lim S. Validation of a wearable cuff-less wristwatch-type blood pressure monitoring device. Sci Rep. 2020 Nov 4;10(1):19015. doi: 10.1038/s41598-020-75892-y. PMID 33149118
- [Background] Muntner P, Shimbo D, Carey RM, Charleston JB, Gaillard T, Misra S, Myers MG, Ogedegbe G, Schwartz JE, Townsend RR, Urbina EM, Viera AJ, White WB, Wright JT Jr. Measurement of Blood Pressure in Humans: A Scientific Statement From the American Heart Association. Hypertension. 2019 May;73(5):e35-e66. doi: 10.1161/HYP.0000000000000087. PMID 30827125
- [Background] Atkinson G, Davison RC, Nevill AM. Performance characteristics of gas analysis systems: what we know and what we need to know. Int J Sports Med. 2005 Feb;26 Suppl 1:S2-10. doi: 10.1055/s-2004-830505. PMID 15702453